CLINICAL TRIAL: NCT00002495
Title: Randomized Trial of Subtotal Nodal Irradiation Versus Doxorubicin, Vinblastine and Subtotal Nodal Irradiation for Stage I-IIA Hodgkin's Disease
Brief Title: SWOG-9133 RT w/ or w/o Doxorubicin and Vinblastine in Stage I or Stage II Hodgkin's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000077691; U10CA032102 (NIH); SWOG-9133 (Other: SWOG); CLB-9391 (Other: CALGB)
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Doxorubicin; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nodal RT (Experimental): subtotal nodal irradiation will consist of mantle and periaortic/spleen fields treated sequentially. Total dose 3600-4000 cGy over 20 fractions.
  Interventions: Radiation: standard subtotal nodal irradiation
- Chemotherapy + Nodal RT (Experimental): 3 cycles (28 days each) of chemotherapy (doxorubicin 25 mg/m^2 on days 1 and 15, vinblastine 6 mg/m^2 on days 1 and 15). Four weeks after last cycle, subtotal nodal irradiation (total dose 3600-4000 cGy over 20 fractions) will be given as described for the Nodal RT arm.
  Interventions: Drug: doxorubicin hydrochloride; Drug: vinblastine; Radiation: standard subtotal nodal irradiation

INTERVENTIONS:
Drug: doxorubicin hydrochloride — 25 mg/m^2 on days 1 and 15
  Arms: Chemotherapy + Nodal RT
Drug: vinblastine — 6 mg/m^2 on days 1 and 15
  Arms: Chemotherapy + Nodal RT
Radiation: standard subtotal nodal irradiation — 3600-4000 cGy delivered over 20 fractions

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with or without doxorubicin and vinblastine in treating patients with stage I or stage II Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare progression-free and overall survival of patients with clinical Stage IA/IIA Hodgkin's disease who have not undergone laparotomy and who are randomized to treatment with subtotal nodal irradiation with vs. without 3 courses of doxorubicin/vinblastine. II. Compare the long-term toxicities associated with these treatments, including cardiopulmonary toxicity, secondary malignancies, and infertility. III. Identify subgroups of patients (based on age, gender, tumor histology, number of disease sites, and presence of high neck presentation) that are particularly responsive to these treatments.

OUTLINE: Randomized study. Arm I: Radiotherapy. Subtotal nodal irradiation using megavoltage equipment (4-10 MeV). Arm II: 2-Drug Combination Chemotherapy followed by Radiotherapy. Doxorubicin, DOX, NSC-123127; Vinblastine, VBL, NSC-49842; followed by subtotal nodal irradiation as in Arm I.

PROJECTED ACCRUAL: 210 patients/arm will be enrolled over about 7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy-proven Hodgkin's disease, subclassified according to the Rye system Clinical Stages IA, IEA, IIA, and IIEA according to modified Ann Arbor system Staging laparotomy not allowed Completely resected disease allowed Residual disease, if present, must be bidimensionally measurable No mediastinal mass greater than 1/3 the maximum chest diameter No infradiaphragmatic presentation No pericardial E lesions (small pericardial effusions in the absence of nodular pericardial disease allowed) Concurrent registration on protocol SWOG-9208 (quality-of-life study) required unless patient does not understand or read English

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: SWOG 0-2 Hematopoietic: AGC at least 2,000 Platelets within normal limits Hepatic: Bilirubin within normal limits Renal: Creatinine within normal limits Cardiovascular: LVEF normal No serious EKG abnormality Pulmonary: No serious pulmonary condition Other: No serious medical condition other than Hodgkin's disease No known AIDS or HIV-associated complex No second malignancy within 5 years except: Adequately treated nonmelanomatous skin cancer Adequately treated in situ carcinoma of the cervix No pregnant or lactating women Adequate contraception required of fertile patients Blood/body fluid analyses to determine eligibility completed within 14 days prior to registration; imaging studies for tumor measurement completed within 28 days prior to registration; screening exams other than blood/body fluid analyses, and imaging studies of nonmeasurable disease or uninvolved organs completed within 42 days prior to registration

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy Chemotherapy: No prior chemotherapy for any reason Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy for any reason Surgery: No staging laparotomy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 1992-09; Primary Completion 2000-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
progression-free survival | every 3 months while on protocol treatment, then every 6 months for 2 years, then annually thereafter
overall survival | every 3 months while on protocol treatment, then every 6 months for 2 years, then annually thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Oliver W. Press, MD, PhD, Study Chair — University of Washington; Todd H. Wasserman, MD, Study Chair — Washington University Siteman Cancer Center
Locations (22):
- United States (22):
  - University of California San Diego Cancer Center, La Jolla, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Ganz PA, Moinpour CM, McCoy S, et al.: Predictors of vitality (energy/fatigue) in early stage Hodgkin's disease (HD): results from Southwest Oncology Group (SWOG) study 9133. [Abstract] J Clin Oncol 22 (Suppl 14): A-6546, 569s, 2004.
- [Result] Ganz PA, Moinpour CM, Pauler DK, Kornblith AB, Gaynor ER, Balcerzak SP, Gatti GS, Erba HP, McCoy S, Press OW, Fisher RI. Health status and quality of life in patients with early-stage Hodgkin's disease treated on Southwest Oncology Group Study 9133. J Clin Oncol. 2003 Sep 15;21(18):3512-9. doi: 10.1200/JCO.2003.01.044. PMID 12972528
- [Result] Press OW, LeBlanc M, Lichter AS, Grogan TM, Unger JM, Wasserman TH, Gaynor ER, Peterson BA, Miller TP, Fisher RI. Phase III randomized intergroup trial of subtotal lymphoid irradiation versus doxorubicin, vinblastine, and subtotal lymphoid irradiation for stage IA to IIA Hodgkin's disease. J Clin Oncol. 2001 Nov 15;19(22):4238-44. doi: 10.1200/JCO.2001.19.22.4238. PMID 11709567
- [Result] Press OW, LeBlanc M, Lichter A, et al.: A phase III randomized intergroup trial of subtotal lymphoid irradiation (STLI) versus doxorubicin, vinblastine, and STLI for stage IA-IIA Hodgkin's disease (SWOG 9133, CALGB 9391). [Abstract] Blood 96(11 pt 1), A-2471, 575a, 2000.